CLINICAL TRIAL: NCT05980078
Title: A Computer-Based Interactive Informed Consent for Surgery Does Not Reduce Decision Conflict
Brief Title: Interactive Informed Consent and Decision Conflict
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor of Surgery and Perioperative Care Department, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017-05-0033
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Upper Extremity Problem

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive consent (Experimental): They were randomized to complete an interactive consent
  Interventions: Other: Interactive consent
- Standard written consent (Active Comparator): They were randomized to complete a standard written consent
  Interventions: Other: Standard consent

INTERVENTIONS:
Other: Interactive consent — They were randomized to complete an interactive consent.
  Arms: Interactive consent
Other: Standard consent — They were randomized to complete a standard written consent.
  Arms: Standard written consent

SUMMARY:
Informed consent for surgery can address the legal aspects while also being simple, informative, and empathic. It can help people confirm that the potential harms are acceptable in light of the potential benefits. Standard consent forms just document this process, while a computer-based, interactive consent process can also standardize and potentially enhance it.

DETAILED DESCRIPTION:
It's not clear that the current informed consent process adequately addresses common misconceptions and adequately confirms patient understanding of potential harms and potential benefits. Thoughtful patient consideration of potential benefits and potential harms of surgery might be facilitated by a step-by-step, iterative, interactive electronic consent process designed to help patients: 1) become aware of their values, 2) understand the actual and potential harms of surgery, 3) understand the potential benefits of surgery, and 4) guide people away from common misconceptions and towards decisions based on their values.

ELIGIBILITY:
Inclusion Criteria:

1. English and Spanish-speaking adults
2. Older than 18 years of age
3. One of six common upper extremity conditions including carpal tunnel release, cubital tunnel release, trigger finger release, plate and screw fixation of a distal radius fracture, removal of a benign lump including a ganglion cyst, and Dupuytren contracture release.

Exclusion Criteria:

People with cognitive deficits were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Decision Conflict Scale | through study completion, an average of 6 months
  The Decision Conflict Scale (DCS) consists of sixteen items rated on a 4-point scale (1 = strongly agree to 4 = strongly disagree), with total scores ranging from 0 to 100. Higher scores indicate greater decisional conflict and therefore a worse outcome.

SECONDARY OUTCOMES:
Jefferson Scale of Patient's Perceptions of Physician Empathy | through study completion, an average of 6 months
  The Jefferson Scale of Patient's Perceptions of Physician Empathy includes five items rated on a 7-point Likert scale (1 = strongly disagree to 7 = strongly agree), with total scores ranging from 5 to 35. Higher scores indicate greater perceived physician empathy, representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Professor of orthopedic surgery at The university of Texas at Austin
Locations (1):
- University of Texas Health Austin (UTHA), Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No